CLINICAL TRIAL: NCT01872559
Title: 3D Sonographic Volumetric Analysis of Ovarian Follicles.
Brief Title: 3 Dimensional Sonography Imaging
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1209013095
Record Dates: First submitted 2013-05-21; First posted 2013-06-07 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: New Imaging Modality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 3D sonographic analysis: The study is designed to evaluate a new imaging modality, 3D sonographic volumetric analysis, and compare it to the conventional 2-dimmensional analysis that is currently in place. Those patients who are scheduled to have an ultrasound as part of their infertility treatment will be offered the opportunity to have additional measurements done at the time of their ultrasound; these additional measurements will take less than 2 minutes and do no require any additional sonograms, tests, or interventions.
  Interventions: Other: 3D Sonography analysis

INTERVENTIONS:
Other: 3D Sonography analysis — Those patients who are scheduled to have an ultrasound as part of their infertility treatment will be offered the opportunity to have additional measurements done at the time of their ultrasound; these additional measurements will take less than 2 minutes and do not require any additional sonograms, tests, or interventions.

SUMMARY:
The study is designed to evaluate a new imaging modality, 3-dimmensional sonographic volumetric analysis, and compare it to the conventional 2-dimmensional analysis that is currently in place. Those patients who are scheduled to have an ultrasound as part of their infertility treatment will be offered the opportunity to have additional measurements done at the time of their ultrasound; these additional measurements will take less than 2 minutes and do no require any additional sonograms, tests, or interventions. All patients are eligible (oocyte donors and autologous oocyte patients) and only patients with a serum estradiol > 2000pg/ML will be enrolled in the study. After the additional measurements are obtained, the results will be digitally stored. The results of the 3D sonographic volumetric analysis will then be correlated with the patients' IVF performance.

DETAILED DESCRIPTION:
The benefits of the study is that 3-dimensional sonographic volumetric analysis may be a superior imaging modality for sonographically assessing oocyte maturity and may lead to change in clinical practice. The lone risk of the study is rooted in protecting the patients' protected health information.

ELIGIBILITY:
Inclusion Criteria:

* All patients (oocyte donors and autologous oocyte patients)with a serum estradiol > 2000pg/ML.

Exclusion Criteria:

* All patients not meeting the estradiol criteria.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: In Vitro fertilization patients and donor egg patients of the Ronald O. Perelman and Claudia Cohen Center for Reproductive Medicine who at the day of monitoring (having an ultrasound and blood work drawn) have an estradiol level greater than 2000pg/ML.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2016-09-16 (Actual)

PRIMARY OUTCOMES:
IVF performance | 3 weeks
  Correlations for age of patient, BMI, documented 2-dimensional sonographic analysis, type of oocyte maturation trigger, serum estradiol prior to trigger, serum estradiol after trigger, number of oocyte retrieved, number of mature oocytes retrieved, embryo grade, type of incubator utilized, day 3 or day 5 transfer, implantation rate, and ultimate pregnancy will be made with the volumetric analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Schattman, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States